CLINICAL TRIAL: NCT03322605
Title: Investigation of the Presence of Residual Tubal Tissue on the Ovarian Surface Following Laparoscopic and Laparotomic Salpingectomy; Do They Really Exist?
Brief Title: Residual Tubal Tissue on the Ovarian Surface Following Salpingectomy With Laparoscopy and Laparotomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Özkan Özdamar, M.D., Istanbul Medeniyet University
Other Study IDs: 2017/250
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Salpingectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Oophorectomy materials during hysterectomy or other gynecological procedures will be examined for fimbrial tissue remnants on their surface
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who undergo salpingo-oophorectomy +/- hysterectomy (laparoscopic or laparotomy) for benign indications, early cervical cancer or low-risk endometrial cancer will be included. Patients with other pelvic malignancies, previous bilateral salpingectomy or bilateral oophorectomy and excessive adhesions will be excluded. Laparoscopy and laparotomy groups will be compared in terms of fibril tissue remnants on the ovarian surface.

DETAILED DESCRIPTION:
Histopathologic data have revealed that up to 70% of ovarian cancers may actually arise from the fallopian tube. Thus, opportunistic bilateral salpingectomy is now promoted for women at the time of hysterectomy for a benign disease. In turn, the potential surgical risks and ovarian cancer prevention of this emerging practice have generated multiple studies, some of which reported microscopic fimbriae were left behind adherent to the ovary. Although it is thought that there is no direct connection between the ovary and its adjacent fallopian tube, the investigators often find remnants of the fimbria adherent to the ovary at the time of surgery. If this tubo-ovarian interface is not separate, then practices such as salpingectomy and radical fimbriectomy may be incomplete, and the effectiveness of this technique as a prophylactic strategy may need reconsideration. In this study, the investigators aim to assess the presence of residual fimbrial/tubal tissue on ovarian surfaces following salpingectomy and to discuss the efficacy of this procedure on the reduction of epithelial ovarian cancer. Patients who undergo salpingo-oophorectomy +/- hysterectomy (laparoscopic or laparotomy) for benign indications, early cervical cancer or low-risk endometrial cancer will be included. Patients with other pelvic malignancies, previous bilateral salpingectomy or bilateral oophorectomy and excessive adhesions will be excluded. Salpingectomy with or without hysterectomy, as indicated, will be performed initially. This will be followed by bilateral oophorectomy as a second step within the same procedure. The ovaries and tubes removed will be sent in separately labelled containers: right tube, left tube, right ovary and left ovary. Histological assessment will be performed by gynecological pathologists. The fallopian tubes will be sectioned serially and ovaries will also be serially sectioned and examined for presence of any remnant tubal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo salpingo-oophorectomy +/- hysterectomy (laparoscopic or laparotomy) for benign indications, early cervical cancer or low-risk endometrial cancer will be included.

Exclusion Criteria:

* Patients with other pelvic malignancies, previous bilateral salpingectomy or bilateral oophorectomy and excessive adhesions will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo salpingo-oophorectomy +/- hysterectomy (laparoscopic or laparotomy) for benign indications, early cervical cancer or low-risk endometrial cancer will be included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of tubal tissue remnants on the ovarian surface | 6 months
  Percentage of tubal tissue remnants on the oophorectomy materials extracted either by laparotomy or laparoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ozkan OZDAMAR, M.D., Principal Investigator — Istanbul Medeniyet University, Faculty of Medicine